CLINICAL TRIAL: NCT02534298
Title: Reorganization of Central Auditory System After Single Sided Deafness: a Functional Magnetic Resonance Imaging Study
Brief Title: Functional Magnetic Resonance Imaging Study of the Central Auditory System After Single Sided Deafness
Acronym: SSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/13/0204; 13 204 02 (Other: University Hospital Toulouse, 2013, DRCI)
Record Dates: First submitted 2015-06-10; First posted 2015-08-27 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Unilateral Hearing Loss
Keywords: single sided deafness.; Auditory plasticity; Asymmetrical hearing loss; Cochlear implants; Inter hemispheric asymmetry; Lateralization index; Dichotic hearing
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single sided deafness (Experimental): single sided deafness and asymmetrical hearing loss patients functional magnetic resonance imaging
  Interventions: Other: functional magnetic resonance imaging
- control group (Other): Normal hearing subject functional magnetic resonance imaging
  Interventions: Other: functional magnetic resonance imaging

INTERVENTIONS:
Other: functional magnetic resonance imaging — functional magnetic resonance imaging

SUMMARY:
The objective is to study the relation between the reorganization of the central auditory system, and the psychophysical deficits in binaural hearing in subjects with single sided deafness.

DETAILED DESCRIPTION:
Background Single sided deafness (SSD) and asymmetrical hearing loss are common hearing impairments, and their social consequences are well established. At the central auditory system level, the single sided deafness is associated with a reorganization of auditory temporal cortices that leads to a reduction of inter hemispheric asymmetry.

Purpose : Our main objective is to study the relation between the reorganization of the central auditory system, namely the inter hemispheric asymmetry, and the psychophysical deficits in binaural hearing in subjects with SSD.

Abstract : Binaural hearing enables spatial localization of the sound source and improves speech recognition in a competing noise. SSD and asymmetrical hearing loss are common hearing impairments, which affect 0.3 to 1/1000 children. In the adult population, this prevalence increases with age. The impact of SSD and asymmetrical hearing loss on quality of life indices is well established and some reports underline its consequences in children scholarship. Previous neuro-imaging and electro physiological studies highlighted the reduction of normal inter hemispheric asymmetry in subjects with SSD. To the best of our knowledge, there is no report about the relation between the central auditory system reorganization and its behavioural deficits.

The investigators propose to conduct a study which analyzes the relationship between the reduction of inter hemispheric asymmetry and performance in binaural hearing tests. Thus, the auditory plasticity will be studied using functional magnetic resonance imaging and more specifically BOLD variations in auditory temporal cortices. A set of binaural hearing assessments will be performed, including speech recognition in noise and localization abilities. The correlation between the lateralization ratio and binaural measurements (speech reception threshold (SRT) in dichotic hearing, diotic hearing, reverse dichotic hearing) will be estimated. Likewise, the impact of SSD duration on cortical reorganization and binaural tests will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed subjects
* SSD confirmed using evoked auditory potentials

Exclusion Criteria:

* Associated neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Lateralization index | 4 weeks
  ratio of the BOLD signal (blood oxygenation level dependent) obtained at the superior temporal cortex in response to stimulation of the monaural sound to the ear BOLD signal obtained for the same stimulus presented binaurally
Speech Reception Threshold | 4 weeks
  signal / noise ratio for the recognition of 50% of the words in dichotic hearing

SECONDARY OUTCOMES:
SRT in reverse dichotic hearing, mean localization error angle | 4 weeks
the percentage of errors in test horizontal location of the sound source | 4 weeks
seniority of deafness | inclusion
  requested information to the patient OR recovered in his medical file

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Marx, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France